CLINICAL TRIAL: NCT05596487
Title: The Effects of End of Life Care Education and Repetitive Standard Patient-Based Simulation on Nursing Students' Knowledge Level, Attitudes and Moods Towards the Patient With Dying Process
Brief Title: The Effect of Repetitive Standardized Patient Simulation and End of Life Care Education on Nursing Students' Knowledge Attitudes and Moods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Betül Çakmak, PHD, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15.03.2021
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: End of Life Care
Keywords: End of life care; standardized patient; nursing; attitude; emotion
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental: repetitive standardized patient simulation (Experimental): In the study, an end-of-life care nursing education program was applied to all students. In the second stage, the standard patient-based practice was performed once with the control group nursing students and twice with the intervention group students.
  Interventions: Other: repetitive standardized patient simulation
- control grup (No Intervention)

INTERVENTIONS:
Other: repetitive standardized patient simulation — In the study, an end-of-life care nursing education program was applied to all students. In the second stage, the standard patient-based practice was performed once with the control group nursing students and twice with the intervention group students. In data collection, an end-of-life care nursing questionnaire, Frommelt attitude scale, positive-negative affect scale, and modified simulation effectiveness tool were used.
  Arms: experimental: repetitive standardized patient simulation

SUMMARY:
This research is a randomized experimental intervention study designed to examine the effect of repetitive standard patient-based education given to nursing students with end-of-life care education nursing on the level of knowledge, attitudes, and moods of the patient's care during the death process.

DETAILED DESCRIPTION:
The research Sample of the study consisted of fourth-year nursing students who agreed to participate in the study (n=50). In the study, an end-of-life care nursing education program was applied to all students. In the second stage, the standard patient-based practice was performed once with the control group nursing students and twice with the intervention group students. In data collection, an end-of-life care nursing questionnaire, Frommelt attitude scale, positive-negative affect scale, and modified simulation effectiveness tool were used.

ELIGIBILITY:
Inclusion Criteria:

* Not having a course in which a four-year undergraduate education is unsuccessful,
* Not participating in the pilot study of the research
* To voluntarily agree to participate in the research.
* Being a fourth-year student in the Department of Nursing

Exclusion Criteria:

* Participating in the pilot study of the research
* Wanting to leave the research.
* Being a first, second and third-year student in the Department of Nursing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-03-19 (Actual)

PRIMARY OUTCOMES:
Knowledge level on end-of-life care nursing | 21 Days
  Evaluated with an end-of-life care nursing questionnaire. This form was developed by the researcher. students answered the test exam. The exam consists of 25 questions. Minimum point is "0" and the maximum point is "100". The higher the score, the higher the knowledge level of the end of life care.
Attitude score toward the care of the patient during the death process | 21 Days
  Evaluated with the scale of Attitude Towards Caring for Dying Patients. Minimum point is "30" and the maximum point is "150". The higher the score, the higher the positive attitude.
positive-negative mood level | 21 Days
  Evaluated with Positive and negative affect:The PANAS Scales-PANAS. It includes 20 emotions, including 10 positive affect and 10 negative affect. It is evaluated in a 5-point Likert type and indicates that the emotion is felt as 1 = very little or not at all, 5 = very much.
evaluate the effectiveness of the simulation environment | 21 Days
  Evaluated with Simulation Effectiveness Tool-Modified. Minimum point is "18" and the maximum point is "95". The higher the score, the higher the positive perception of the learning activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No